CLINICAL TRIAL: NCT06801002
Title: A Phase 1, Open-label, Dose-escalation and Expansion, First-in-human Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of JBZ-001, a Dihydroorotate Dehydrogenase (DHODH) Inhibitor, in Patients With Advanced Solid and Hematological Malignancies
Brief Title: Trial to Evaluate the Safety & Tolerability of JBZ-001 in Pts With Advanced Solid and Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jabez Bioscience, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JBZ-001-101
Record Dates: First submitted 2024-11-07; First posted 2025-01-30 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; lymphoma; NHL; Non-Hodgkin's lymphoma; DHODH; Small Molecule; DHO
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Experimental Cohort 1 (Experimental): 1~6 subjects in this cohort will receive 1 dose 5 mg orally.
  Interventions: Drug: JBZ-001
- Experimental Cohort 2 (Experimental): 1~6 subjects in this cohort will receive 1 dose 5 mg orally daily
  Interventions: Drug: JBZ-001
- Experimental Cohort 3 (Experimental): 1~6 subjects in this cohort will receive 1 dose of 10 mg orally daily
  Interventions: Drug: JBZ-001
- Experimental Cohort 4 (Experimental): 1~6 subjects in this cohort will receive 1 dose of 17.5 mg orally daily
  Interventions: Drug: JBZ-001
- Experimental Cohort 5 (Experimental): 1~6 subjects in this cohort will receive 1 dose of 25 mg orally daily
  Interventions: Drug: JBZ-001

INTERVENTIONS:
Drug: JBZ-001 — JBZ-001 Oral Capsule

SUMMARY:
This will be a phase 1, open-label, dose-escalation and expansion, FIH trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of JBZ-001, a DHODH inhibitor, in patients with refractory solid and hematological malignancies. The study design includes two independent parts: dose escalation in solid tumors and NHL (Part 1), and up to four indication expansions in selected solid tumor types and NHL (Part 2). The dose escalation will enroll patients with solid tumors and NHL following a standard "3+3" design enrolling a minimum of 3 and up to 6 patients per dose level.

DETAILED DESCRIPTION:
This will be a phase 1, open-label, dose-escalation and expansion, FIH trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of JBZ-001, a DHODH inhibitor, in patients with refractory solid and hematological malignancies. The study will enroll patients with solid tumors and NHL. The study design includes two independent parts: dose escalation in solid tumors and NHL (Part 1), and up to four indication expansions in selected solid tumor types and NHL (Part 2). The dose escalation will enroll patients with solid tumors and NHL following a standard "3+3" design enrolling a minimum of 3 and up to 6 patients per dose level. Single-patient efficacy signals (i.e. CR or PR) may be followed in an efficacy-signal dose expansion cohort of up to 10 patients on any given dose level with the same tumor type. In addition to dose-limiting toxicity (DLT) evaluation during dose escalation, a Bayesian safety monitoring rule will be used to evaluate the rate of DLTs during cohort expansions. The study includes subgroup-specific eligibility criteria, DLTs, safety and efficacy monitoring, and other indication-relevant aspects. Patients with clinical benefit may be treated until disease progression or toxicity.

The primary objective is to evaluate the safety and tolerability and establish an OBD of single agent JBZ-001 in patients with solid tumors and NHL. Secondary objectives include efficacy endpoints and the PK of single agent JBZ-001. To characterize the JBZ-001 single dose PK profile, the patients enrolled in the first dose level will first receive a single dose of JBZ-001 followed by one-week off-drug (Cycle 0). Exploratory objectives include correlative studies of plasma cell expression of CD38, CD47, and other markers.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age, at the time of signing the informed consent.
2. Dose escalation and expansion:

   1. Solid tumors: have a histologically confirmed relapsed or refractory advanced solid tumor for which no standard approved treatment is available, or is ineligible for, or did not tolerate standard approved treatment.
   2. NHL: have a histologically confirmed relapsed or refractory diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL) or Mantle cell lymphoma (MCL) for which no standard approved treatment is available, or is ineligible for, or did not tolerate standard approved treatment.
3. Measurable/evaluable disease or documented relapse, respectively, relevant for tumor type as follows:

   1. Solid tumors: per Response evaluation criteria in solid tumors (RECIST) 1.1 with at least one target lesion
   2. NHL: Measurable disease defined as ≥1 measurable nodal lesion (long axis >1.5 cm and short axis >1.0 cm) or ≥1 measurable extra-nodal lesion (long axis >1.0 cm) on computed tomography (CT) scan or magnetic resonance imaging (MRI)
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. All previous anti-cancer therapy-related AEs should have resolved to grade 1 or baseline value with the exception of alopecia and stable, treated endocrine toxicities of immune checkpoint inhibitors (ICIs) Note: Subjects with irreversible toxicity that in the opinion of the treating physician is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, hormone deficiency requiring replacement therapy) -

Exclusion Criteria:

1. Known hypersensitivity to JBZ-001 or any of its excipients
2. Corrected interval between Q and T wave on ECG (QTc) ≥ 470 msec using Fredericia's formula.
3. Has significant and symptomatic cardiovascular disease (such as congestive heart failure New York Heart Association class III or higher, myocardial infarction, cerebrovascular disease, unstable angina, unstable arrhythmia) within the 3 months prior to first dose of JBZ-001.
4. Has another malignant disease requiring treatment, with the exception of curatively treated malignancies or malignancies with very low potential for recurrence or progression.
5. For solid tumor subjects:

   1. Symptomatic ascites or pleural effusion. A subject who is clinically stable for 2 weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
   2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks prior to study entry, as long as the dose is ≤ 4 mg of dexamethasone or equivalent per day
6. Known active HIV infection on antiretroviral therapy. Note: Testing is not required for eligibility.
7. Known active infection with hepatitis B or hepatitis C. Note: Testing is not required for eligibility.
8. Any other active infection requiring systemic therapy.
9. Major surgery (excluding procedures to stabilize the vertebrae) within 4 weeks or minor surgery within 2 weeks prior to first dose of JBZ-001.
10. Has a history of GI surgery or other procedures that might interfere with the absorption or swallowing of the study drug.
11. History or clinical evidence of any medical condition which the investigator judges as likely to interfere with the results of the study, poses an additional risk in participating, or makes the subject unlikely to comply with the study-related visits and assessments.
12. Female participants: pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all adverse events | 28 Days
  Evaluation of adverse events
Maximum tolerated dose (MTD） | 28 days
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 33days of multiple dosing.
Phase II dose (RP2D) | 28 days
  The number and proportion of patients experiencing at least 1 dose-limiting toxicity (DLT) will be used as the primary measure to evaluate the RP2D

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax） | 28 days
  Pharmacokinetic (PK) parameters after a single oral dose & multiple doses
Time to Cmax (tmax) | 28 days
  Pharmacokinetic (PK) parameters after a single oral dose & multiple doses
Area under the serum concentration-time curve (AUC[0-t] | 28 days
  Pharmacokinetic (PK) parameters after a single oral dose & multiple doses
Area under the serum concentration-infinity curve AUC[0-infinity] | 28 days
  Pharmacokinetic (PK) parameters after a single oral dose & multiple doses
Apparent terminal phase half-life (t1/2) | 28 days
  Pharmacokinetic (PK) parameters after a single oral dose
Overall Response Rate (ORR) | up to 1 year(anticipated)
  The proportion of patients with complete response (CR) and partial response (PR)
Duration of response (DoR) | up to 1 year(anticipated)
  The time from the date when the measurement criteria were met for complete or partial response (whichever occurred first) until the date of the first observed Progression Disease or death as a result of any cause.
Progression-free survival (PFS) | up to 1 year(anticipated)
  The time the patient is enrolled to the date of any recorded disease progression or the death of any cause.
Time to Progression (TTP) | up to 1 year(anticipated)
  The time from clinical remission to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Jirakova, MD PhD, Study Chair — Jabez Biosciences, Inc
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: Undecided